CLINICAL TRIAL: NCT05607459
Title: Efficacy of Adding Dry Needling to a Manual Therapy and Therapeutic Exercise Interventions for Managing Neck Pain Populations: A Randomized Controlled Trial
Brief Title: Dry Needling, Manual Therapy and Exercise for Neck Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Ortiz, Vice-dean of research, Camilo Jose Cela University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhD-MML
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain, Posterior
Keywords: Dry Needling
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, controlled and single-blinded clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): This group will receive dry needling, manual therapy (consisting of a manual compression over myofascial trigger points located at the upper trapezius muscle, scalene muscles and cervical multifidus) and therapeutic exercise interventions
  Interventions: Other: Dry Needling; Behavioral: Therapeutic Exercise; Other: Manual Therapy
- Sham Dry Needling Group (Active Comparator): This group will receive manual therapy (consisting of a manual compression over myofascial trigger points located at the upper trapezius muscle, scalene muscles and cervical multifidus), therapeutic exercise interventions and a previously described sham dry needling intervention.
  Interventions: Behavioral: Therapeutic Exercise; Other: Manual Therapy; Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry Needling — Dry needling consists of a skilled intervention which uses a thin filiform needle (as those used in acupuncture) to penetrate the skin and stimulate underlying myofascial trigger points (defined as "a hyperirritable spot in skeletal muscle that is associated with a hypersensitive palpable nodule in a taut band which is painful on manual compression and can give rise to characteristic referred pain, referred tenderness, motor dysfunction and autonomic phenomena.")
  This intervention will be performed targeting the upper trapezius and cervical multifidus muscles
  Arms: Dry Needling Group
Behavioral: Therapeutic Exercise — Patients will include a supervised therapeutic exercise program in their daily life, based on strengthening exercises for neck muscles.
Other: Manual Therapy — Patients will receive a manual compression (30 seconds) over myofascial trigger points located at the upper trapezius muscle, scalene muscles and cervical multifidus muscle.
Other: Sham Dry Needling — For the sham DN intervention, a similar approach will be used, but the skin will be not pierced since the material used will be a telescopic Park's sham device.
  The guide tube will be pressed against the skin mark and the sham needle will be allowed to drop. The handle will be tapped briskly, but the (blunted) needle tip will not not break the skin.
  Arms: Sham Dry Needling Group

SUMMARY:
Since neck pain is the fourth highest disabling condition (with an estimated point prevalence of 20%, lifetime prevalence up to 70% and high recurrence rates), dry needling targeting myofascial trigger points in neck muscles has been proposed as an effective treatment for reducing pain and disability in patients with chronic neck pain.

A recent meta-analysis reported whether dry needling could be recommended for this population. Low to moderate evidence suggests that dry needling can be effective at the short-term, but its effects on pressure pain sensitivity or cervical range of motion are limited.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18 and 65 years old
* To have been experiencing unilateral neck pain for at least 3 months
* To have a Neck Disability Index (NDI) score >8
* To have a Visual Analogue Scale (VAS) score >3
* To have at least one active MTrP located in the upper trapezius or cervical multifidus muscles

Exclusion Criteria:

* History of whiplash injury
* Previous cervical surgery
* Cervical radiculopathy or myelopathy
* Diagnosis of fibromyalgia
* Additional analgesic treatments during the study (e.g. physiotherapy or drugs)
* Psychiatric disorders
* Any contraindication to the interventions proposed (e.g. fear of needles or anticoagulants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  A 100mm visual analogue scale will be used. The patient will indicate the level of pain intensity from 0 (no pain) to 10 (the worst pain imaginable)
Visual Analogue Scale | One month follow-up
  A 100mm visual analogue scale will be used. The patient will indicate the level of pain intensity from 0 (no pain) to 10 (the worst pain imaginable)
Visual Analogue Scale | Three months follow-up
  A 100mm visual analogue scale will be used. The patient will indicate the level of pain intensity from 0 (no pain) to 10 (the worst pain imaginable)
Visual Analogue Scale | Six months follow-up
  A 100mm visual analogue scale will be used. The patient will indicate the level of pain intensity from 0 (no pain) to 10 (the worst pain imaginable)
Visual Analogue Scale | Twelve months follow-up
  A 100mm visual analogue scale will be used. The patient will indicate the level of pain intensity from 0 (no pain) to 10 (the worst pain imaginable)

SECONDARY OUTCOMES:
Pittsburg Sleeping Quality Index | Baseline
  This is a validated self-reported questionnaire assessing the sleeping quality. Scores range from 0 (best sleep quality) to 21 (worst sleep quality)
Pittsburg Sleeping Quality Index | One month follow-up
  This is a validated self-reported questionnaire assessing the sleeping quality. Scores range from 0 (best sleep quality) to 21 (worst sleep quality)
Pittsburg Sleeping Quality Index | Three months follow-up
  This is a validated self-reported questionnaire assessing the sleeping quality. Scores range from 0 (best sleep quality) to 21 (worst sleep quality)
Pittsburg Sleeping Quality Index | Six months follow-up
  This is a validated self-reported questionnaire assessing the sleeping quality. Scores range from 0 (best sleep quality) to 21 (worst sleep quality)
Pittsburg Sleeping Quality Index | Twelve months follow-up
  This is a validated self-reported questionnaire assessing the sleeping quality. Scores range from 0 (best sleep quality) to 21 (worst sleep quality)
Hospital Anxiety and Depression Scale | Baseline
  This is a validated self-reported questionnaire assessing the level of anxiety and depression in two subscales (HADS-A and HADS-D). Scores for each scale range from 0 to 21 points, where lower scores are associated with lower depressive and anxiety levels.
Hospital Anxiety and Depression Scale | One month follow-up
  This is a validated self-reported questionnaire assessing the level of anxiety and depression in two subscales (HADS-A and HADS-D). Scores for each scale range from 0 to 21 points, where lower scores are associated with lower depressive and anxiety levels.
Hospital Anxiety and Depression Scale | Three months follow-up
  This is a validated self-reported questionnaire assessing the level of anxiety and depression in two subscales (HADS-A and HADS-D). Scores for each scale range from 0 to 21 points, where lower scores are associated with lower depressive and anxiety levels.
Hospital Anxiety and Depression Scale | Six months follow-up
  This is a validated self-reported questionnaire assessing the level of anxiety and depression in two subscales (HADS-A and HADS-D). Scores for each scale range from 0 to 21 points, where lower scores are associated with lower depressive and anxiety levels.
Hospital Anxiety and Depression Scale | Twelve months follow-up
  This is a validated self-reported questionnaire assessing the level of anxiety and depression in two subscales (HADS-A and HADS-D). Scores for each scale range from 0 to 21 points, where lower scores are associated with lower depressive and anxiety levels.
Neck Disability Index | Baseline
  This is a validated self-reported questionnaire assessing the neck pain disability. Scores range from 0 (absence of disability) to 100 (worst disability).
Neck Disability Index | One month follow-up
  This is a validated self-reported questionnaire assessing the neck pain disability. Scores range from 0 (absence of disability) to 100 (worst disability).
Neck Disability Index | Three months follow-up
  This is a validated self-reported questionnaire assessing the neck pain disability. Scores range from 0 (absence of disability) to 100 (worst disability).
Neck Disability Index | Six months follow-up
  This is a validated self-reported questionnaire assessing the neck pain disability. Scores range from 0 (absence of disability) to 100 (worst disability).
Neck Disability Index | Twelve months follow-up
  This is a validated self-reported questionnaire assessing the neck pain disability. Scores range from 0 (absence of disability) to 100 (worst disability).
Tampa Scale for Kinesiophobia | Baseline
  The scale consist of 11 items where patients have to choose in a 4-point Likert scale how much they agree with each item, being 1 "complete disagreement" and 4 "complete agreement" (total score from 0 to 44), where higher scores indicate greater kinesiophobia.
Tampa Scale for Kinesiophobia | One month follow-up
  The scale consist of 11 items where patients have to choose in a 4-point Likert scale how much they agree with each item, being 1 "complete disagreement" and 4 "complete agreement" (total score from 0 to 44), where higher scores indicate greater kinesiophobia.
Tampa Scale for Kinesiophobia | Three months follow-up
  The scale consist of 11 items where patients have to choose in a 4-point Likert scale how much they agree with each item, being 1 "complete disagreement" and 4 "complete agreement" (total score from 0 to 44), where higher scores indicate greater kinesiophobia.
Tampa Scale for Kinesiophobia | Six months follow-up
  The scale consist of 11 items where patients have to choose in a 4-point Likert scale how much they agree with each item, being 1 "complete disagreement" and 4 "complete agreement" (total score from 0 to 44), where higher scores indicate greater kinesiophobia.
Tampa Scale for Kinesiophobia | Twelve months follow-up
  The scale consist of 11 items where patients have to choose in a 4-point Likert scale how much they agree with each item, being 1 "complete disagreement" and 4 "complete agreement" (total score from 0 to 44), where higher scores indicate greater kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera Calero, PhD, Principal Investigator — Camilo José Cela University
Locations (1):
- Juan Antonio Valera-Calero, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No